CLINICAL TRIAL: NCT05302986
Title: Benefits on Post-operative Pain of Intravenous, Intraoperative, Tranexamic Acid Injection During Arthroscopic Shoulder Surgery.
Brief Title: Effect on Post-operative Pain of Tranexamic Acid Injection During Shoulder Surgery
Acronym: ASCOT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASCOT; 2021-005710-34 (Other: ANSM)
Record Dates: First submitted 2022-03-02; First posted 2022-03-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Disease
Keywords: Shoulder; Pain; Arthroscopic shoulder surgery
MeSH Terms: conditions — Pain | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, national monocentric study, randomized in parallel groups, comparative versus placebo, double-blind (patient and investigating surgeon).
  * Group 1: Surgery with intravenous injection of tranexamic acid
  * Group 2: Surgery with intravenous injection of Placebo (0.9% sodium chloride)
Who Masked: Participant, Investigator
Masking Description: The study will be conducted in a double-blind setting. The patient and the investigating surgeon will be blinded. The injection of the product will be performed by the anesthetist that will be aware of the injected product (tranexamic acid or sodium chloride).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery with intravenous injection of tranexamic acid (Experimental): The dose will be 0.1 mg / kg (= 10 mg/kg) and diluted in a 100 mL infusion bag of sodium chloride. The product will have to be administered as a slow infusion over 10 minutes.
  Interventions: Drug: Tranexamic acid injection
- Surgery with intravenous injection of Placebo (0.9% sodium chloride) (Placebo Comparator): A 100 mL infusion bag of sodium chloride will be administered as a slow infusion over 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid injection — The dose will be 0.1 mg / kg (= 10 mg/kg) and diluted in a 100 mL infusion bag of sodium chloride. The product will have to be administered as a slow infusion over 10 minutes during the shoulder surgery.
  Arms: Surgery with intravenous injection of tranexamic acid
Drug: Placebo — Surgery with intravenous injection of Placebo (0.9% sodium chloride). A 100 mL infusion bag of sodium chloride will be administered as a slow infusion over 10 minutes during shoulder surgery.
  Arms: Surgery with intravenous injection of Placebo (0.9% sodium chloride)

SUMMARY:
Arthroscopic shoulder surgery is a commonly performed minimally invasive surgery in which a camera (an arthroscope) is inserted inside the shoulder joint.

This surgery is responsible for moderate to severe pain. It may require the use of opioid analgesics in the acute phase. One of the components of this pain may be the postoperative hematoma.

Pain is one of the main causes of patient satisfaction failure after shoulder surgery. Finding ways to reduce this pain is a primary principle in the management of this surgery. Until now, this management requires the frequent use of morphine. However, this use of morphine may conduct to adverse effects (nausea/vomiting, constipation, malaise, sweating), and even public health problems such as addiction.

It is therefore interesting to look for ways to increase the patient's analgesia by other means, which will thus increase patient satisfaction and make his management more fluid. The effect on pain of hematoma reduction is rarely described in the scientific literature.

The hypothesis of this study is that the intraoperative administration of intravenous (IV) tranexamic acid can reduce the hematoma and thus decrease postoperative pain.The aim of this study is to demonstrate that the use of IV tranexamic acid intraoperatively, compared to a placebo (sodium chloride 0.9%), reduces postoperative pain after arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

1 - Male or female aged 18 years old or more; 2- Patient requiring shoulder arthroscopy; 3 - Patient affiliated to a social security scheme; 4 - Patient informed on the study and who has signed the informed consent form.

Exclusion Criteria:

1. - Tranexamic acid contraindications (Hypersensitivity to the active substance or to any of the excipients, Acute venous or arterial thrombosis, Severe renal impairment, History of convulsions);
2. - Pregnant or breastfeeding patient;
3. - Patient under legal protection;
4. - Patient taking part simultaneously to another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the use of morphine treatments in the 24 postoperative hours (yes/no). | At 24 hours post-operative
  Evaluation of the use of morphine treatments in the 24 postoperative hours (yes/no).

SECONDARY OUTCOMES:
Evaluation of postoperative shoulder pain between the two groups | At 24 hours and 7 days after surgery
  Shoulder pain is assessed through a Visual Analog Scale (0-100) performed 24 hours post-operative and 7 days after surgery (online assessment with the help of software)
Evaluation of patient satisfaction between the two groups | The day after surgery
  Satisfaction will be assessed through an Evaluation of the Experience of General Anesthesia questionnaire.
Assessment of shoulder functionality between the two groups | Before surgery and at the day 30 after surgery
  The functionality of the shoulder will be evaluated by the Subjective Shoulder Value scale.
  Not normal shoulder that would scored 0% and normal shoulder that would scored 100%.
Assessment of shoulder functionality between the two groups | Before surgery and at the day 30 after surgery
  The functionality of the shoulder will be evaluated by the Constant Score.
Evaluation of the safety of the treatments under study between the two groups | Continuously from surgery up to 30 days after surgery
  Collection of adverse events throughout the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Jean Villar, Bruges, France, France

REFERENCES:
- [Background] Hartland AW, Teoh KH, Rashid MS. Clinical Effectiveness of Intraoperative Tranexamic Acid Use in Shoulder Surgery: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Sep;49(11):3145-3154. doi: 10.1177/0363546520981679. Epub 2021 Jan 21. PMID 33475421
- [Background] Chevet I, Remerand F, Couvret C, Baud A, Pouplard C, Rosset P, Laffon M, Fusciardi J. [Tranexamic acid reduces haematomas but not pain after total knee arthroplasty]. Ann Fr Anesth Reanim. 2011 Jan;30(1):17-24. doi: 10.1016/j.annfar.2010.11.017. Epub 2011 Jan 6. French. PMID 21215592
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Liu YF, Hong CK, Hsu KL, Kuan FC, Chen Y, Yeh ML, Su WR. Intravenous Administration of Tranexamic Acid Significantly Improved Clarity of the Visual Field in Arthroscopic Shoulder Surgery. A Prospective, Double-Blind, and Randomized Controlled Trial. Arthroscopy. 2020 Mar;36(3):640-647. doi: 10.1016/j.arthro.2019.10.020. Epub 2019 Dec 20. PMID 31870749
- See also: Tranexamic acid (TXA) is widely used across surgical specialties to reduce perioperative bleeding. — https://pubmed.ncbi.nlm.nih.gov/33475421/
- See also: Tranexamic acid (TxA) reduces total blood losses (TBL) and allogenic transfusion (TH) after total knee arthroplasty (TKA). — https://pubmed.ncbi.nlm.nih.gov/21215592/
- See also: Several methods have been devised to estimate shoulder function. — https://pubmed.ncbi.nlm.nih.gov/3791738/
- See also: To determine whether intravenous administration of tranexamic acid (TXA) before shoulder arthroscopic rotator cuff repair surgery can improve arthroscopy visual clarity. — https://pubmed.ncbi.nlm.nih.gov/31870749/